CLINICAL TRIAL: NCT00394680
Title: Stents, Drug Eluting Stents, and CABG- Financial and Clinical Impact.
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Other Study IDs: CABGvsStent-Jerusalem
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Coronary Arteriosclerosis; Angina Unstable; Myocardial Infarction
Keywords: coronary revascularization; stent inmplantation; coronary bypass
MeSH Terms: conditions — Coronary Artery Disease; Angina, Unstable; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Options for coronary revascularization include stent implantation and coronary bypass surgery. Both modalities have their unique advantages and disadvantages in terms of clinical outcomes as well as financial impact on the medical system. We wish to investigate the late results of patients undergoing coronary revascularization, the need for re-hospitalization, re-intervention, patient satisfaction as well as the financial burden on the medical system. The study will be conducted by historical prospective review of hospital records in conjunction with records of the medical insurance companies ("HMO's").

DETAILED DESCRIPTION:
Cardio-vascular disease is the second leading cause of death in the western world. Two modes of treatment are currently used:

Coronary Artery Bypass Graft (CABG) Percutaneous Interventions (PCIs) i.e: balloon angioplasty and stents[ bare metal (BMS) and drug eluting (DES)].

CABG is a major operation but is considered to be safe and with good quality of life in the years to follow. The initial cost of CABG is high but usually stays low thereafter.

PCI is less invasive but its downfall is a high rate of restenosis hence leading to the return of angina. The initial cost is low but due to the return of symptoms the cost increases.

The goal of DES is to lower the rate of restenosis thus reducing the need for repeat hospitalizations and procedures. The initial cost of this stent is higher than that of the BMS but still lower than that of CABG.

The goal of this study is to assess and compare the average annual cost of treatment for patients with multi-vessel disease who underwent one of the following procedures:

1. CABG
2. DES
3. BMS

The information for the study is derived from the data bases of the cardiology and cardio-thoracic surgery departments at Shaarey-Zedek hospital and from those of Clalit Health Services and Kupat Holim Meuhedet.

The study design is historical prospective. The participants are insured by the above mentioned HMOs and were treated during 2000-2004.

The final sample's size will be decided on according to a pilot study with 15 patients from each of the treatment groups.

To our knowledge no studies comparing CABG and DES have yet been published. We believe that our study could become a mile stone in the process of choosing the most suitable treatment for the patient and for the health system.

ELIGIBILITY:
Inclusion Criteria:

* Patients which are insured in the relevant HMO's and suffer from a multi-vessel coronary disease with occlusion of at least 70% of at least two of the main coronary vessels.

Exclusion Criteria:

* Non multi- vessel Disease
* Any additional cardiac disease

  1. Valvular
  2. Low EF (<30%)
* Liver disease - according to liver enzymes
* Other cardiac treatment (past or immediate future)

  1. Active MI (24hrs before revascularization)
  2. Previous revascularization before beginning of follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients which are insured in the relevant HMO's and suffer from a multi-vessel coronary disease and were treated during 2000-2004
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2006-11; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Shmueli, PhD, Principal Investigator — The Hebrew University, School of Public Health